CLINICAL TRIAL: NCT02126371
Title: LP0058-1005 - A Phase I, Open-Label, Four-Way Crossover and Food-Effect Study of LEO 32731 in Healthy Subjects When Administered as an Immediate and Modified Release Formulation
Brief Title: LP0058-1005 - A Open-Label, Four-Way Crossover and Food-Effect Study of LEO 32731 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: LP0058-1005
Record Dates: First submitted 2014-04-07; First posted 2014-04-30 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Other): LEO32731
  Interventions: Drug: LEO32731

INTERVENTIONS:
Drug: LEO32731

SUMMARY:
LEO 32731 ("Study Drug") is an investigational drug which is being developed by LEO Pharma A/S ("the Sponsor"), with an aim to help people with skin conditions called psoriasis. The aim (s) of this Study are to determine:

* The effects of the Study Drug when given as different formulations intended for oral administration (tablets and capsules)
* The safety of the Study Drug and any side effects that might be associated with it
* The effect of food on the Study Drug
* The Study will also measure how much of the Study Drug gets into the blood stream and how long it takes the body to remove it and what affect the Study Drug has on the body.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be males of any ethnic origin between 18 and 55 years of age
2. Subjects will have a body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive
3. Subjects must be in good health, as determined by: a medical history, physical examination, vital sign assessment, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations (congenital non haemolytic hyperbilirubinaemia is NOT acceptable)
4. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions

Exclusion Criteria:

1. Male subjects who are not willing, or whose partners are not willing, to use appropriate contraception (such as a condom with spermicidal foam/gel/film/cream/suppository), or donate sperm from the time of the first dose until 3 months after the final dosing occasion. Male subjects whose partners are of child-bearing potential must also agree to use an additional highly effective method of contraception
2. Subjects who have an abnormality in heart rate, blood pressure, temperature or respiration rate that, in the opinion of the investigator, increases the risk of participating in the study, in accordance with Covance current reference ranges at screening confirmed by a repeat assessment.
3. Subjects who have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risk of participating in the study, confirmed by a repeat ECG: such as QTcB interval >450 msec, 2nd or 3rd degree, Atrioventricular block, complete left bundle branch block, complete right bundle branch block, Wolff-Parkinson-White Syndrome, defined as PR<110 msec,
4. Subjects who have received: any prescribed systemic or topical medication within 14 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety. slow release medicinal formulations considered to still be active within 14 days of the first dose administration, unless in the opinion of the Investigator, the medication will not interfere with the study procedures or compromise safety.
5. Subjects who are still participating in a clinical study (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical entity) in the past 3 months prior to the first dosing occasion
6. Subjects with a significant history of drug allergy as determined by the Investigator.
7. Subjects who have any clinically significant allergic disease (excluding non-active hayfever) as determined by the Investigator.
8. Subjects with, or with a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological or other major disorders as determined by the Investigator.
9. Subjects who: are known to have serum hepatitis, are carriers of the hepatitis B surface antigen (HBsAg) are carriers of the hepatitis C antibody, have a positive result to the test for HIV antibodies, have a history of active tuberculosis or history of incompletely treated tuberculosis within the last 5 years, confirmed by their medical records

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | one week

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | one week

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Brooks, MD, Principal Investigator — Covance CRU
Locations (1):
- Covance CRU, Leeds, United Kingdom